CLINICAL TRIAL: NCT05510882
Title: Effects of Different Treatment Modalities for Obstructive Sleep Apnea on Temporomandibular Joint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: not sponsered
Record Dates: First submitted 2022-08-08; First posted 2022-08-22 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2022-08

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; tempromandibular joint
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- three groups of different treatment modalities for OSA (Other): Group I: patients were treated with CPAP. Group II: patients were treated with digitally fabricated MAD. Group iII: patients were treated with oral myofunctional therapy.
  Interventions: Other: different treatment modalities for OSA

INTERVENTIONS:
Other: different treatment modalities for OSA — Group I: patients will be treated with CPAP. Group II: patients will be treated with digitally fabricated MAD. Group II: patients will be treated with physical therapy.
  Other Names: treatment

SUMMARY:
this study aims to evaluate the subjective symptoms, clinical and radiographic signs of temporomandibular disorders related to the use of CPAP, MAD and physical therapy in the treatment of patients with obstructive sleep apnea.

DETAILED DESCRIPTION:
The study will be conducted on thirty-nine patients with OSA attending to sleep disorders breathing Unit, Chest Department at Mansoura University Hospital confirmed by polysomnography in the period between July and September 2022. The patients will be divided equally into three therapy groups each compromise 13 patients:

Group I: patients will be treated with CPAP. Group II: patients will be treated with digitally fabricated MAD. Group II: patients will be treated with physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* • All adult patients, diagnosed as having OSA after full night polysomnography.

Exclusion Criteria:

* • Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
This study aims to assess signs of temporomandibular disorders related to the use of CPAP, MAD and physical therapy in the treatment of patients with OSA. | up to four months
  Pain scoring will be measured through a visual analogue scale (VAS) with 0 scores for no pain and 10 scores for worst pain experien Clicking was assessed as to its presence=1 or absence=0 The maximal unassisted, pain-free mouth opening will be measured in millimeters using a Vernier caliper Lateral movements: will be measured as the horizontal distance extending from maxillary midline to mandibular midline in millimeters using Vernier caliper All measurements record will be considered as a baseline to be used in comparison with 3 months post-treatment records

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No
The study will be conducted on thirty-nine patients with OSA attending to sleep disorders breathing Unit, Chest Department at Mansoura University Hospital confirmed by polysomnography in the period between July and September 2022.

REFERENCES:
- [Derived] Attia AAMM, Awad SS, Mansour M, Baz H, Zahran KM, Saleh AM. Effects of different treatments for obstructive sleep apnea on temporomandibular joint: a randomized clinical trial. BMC Oral Health. 2024 Aug 11;24(1):931. doi: 10.1186/s12903-024-04623-w. PMID 39129005